CLINICAL TRIAL: NCT03222531
Title: Expanding the Pool in Orthotopic Heart Transplantation: The Use of Hepatitis C Positive Donor Hearts in Hepatitis C Negative Recipients
Brief Title: Expanding the Pool in Orthotopic Heart Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mary E. Keebler, MD (Other)
Responsible Party: Sponsor-Investigator, Mary E. Keebler, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19030424
Record Dates: First submitted 2017-07-05; First posted 2017-07-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C; Heart Transplant; Cardiac Transplant
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV seropositive non-viremic (HCV Ab+/NAT-) donor (Experimental): HCV seropositive non-viremic (HCV Ab+/NAT-) donor hearts to HCV seronegative recipients.
  Heart recipients will be monitored for HCV for one year following transplant. When HCV RNA is detected, the transmission-triggered treatment phase will be initiated.
  Recipients will be treated with 12-week oral course of sofosbuvir/velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
  Intervention: Drug: sofosbuvir/velpatasvir
  Interventions: Drug: sofosbuvir/velpatasvir
- HCV seropositive viremic (HCV Ab+/NAT+) donor (Experimental): HCV seropositive viremic (HCV Ab+/NAT+) donor hearts to HCV seronegative recipients.
  Starting post-operative day 1, heart recipients will be treated with 12-week oral course of sofosbuvir/velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
  Intervention: Drug: sofosbuvir/velpatasvir
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — Drug: sofobuvir/velpatasvir
  Other Names: Epclusa

SUMMARY:
This is an open-label, pilot trial to test the safety and efficacy of transplantation of hearts from HCV seropositive non-viremic (HCV Ab+/NAT-) and HCV seropositive viremic (HCV Ab+/NAT+) donors to HCV seronegative recipients on the heart transplant waitlist. Treatment and prophylaxis will be administered, using a transmission-triggered approach for the first scenario (HCV Ab+/NAT- donors, arm 1) and a prophylaxis approach for the later scenario (HCV Ab+/NAT+ donors, arm 2).

DETAILED DESCRIPTION:
This is a prospective, single center, pilot, open-label study of transplantation of hearts of HCVAb+ donors to HCVAb- recipients with subsequent therapy with sofosbuvir/velpatasvir (Epclusa®). Recipients of a heart from HCVAb+/NAT- donors is ARM 1 or the transmission-triggered arm of the study. In this arm, the study will monitor transmission of HCV by measuring HCV RNA in heart transplant recipients. If HCV RNA is detected, indicating transmission of HCV, recipients will be treated with sofosbuvir/velpatasvir (Epclusa®) for 12 weeks. Virological response will be assessed at 4 weeks, end of treatment and 12 weeks after completion of therapy.

Recipients of a heart from HCVAb+/NAT+ donors will be in ARM 2 or the prophylaxis arm of the study. In this arm, patients will be started on a 12-week course of sofosbuvir/velpatasvir (Epclusa®) on post-operative day 1 and will undergo close monitoring of HCV RNA for evidence of transmission as well as monitoring of adverse events from therapy.

ELIGIBILITY:
Inclusion criteria (recipients):

* End stage heart failure
* Age ≥ 18 and <71 years
* Listed heart transplant at UPMC
* Have panel reactive antibody level of <98%
* No obvious contraindication to liver transplant
* Able to travel to UPMC for routine post-transplant visits and study visits for a minimum of 12 months after transplantation
* Able to provide informed consent
* Be willing to use a contraceptive method for a year after transplant

Inclusion criteria (donors):

* HCV antibody positive
* HCV NAT negative or positive
* Acceptable cardiac function for donation

Exclusion criteria (recipients):

* HIV positive
* HCVAb or HCV RNA positive
* Presence of behavioral risk factors for contracting HCV. These behavioral risk factors are current injection drug use, current intranasal illicit drug use, current percutaneous/parenteral exposures in an unregulated setting.
* Hepatitis B surface antigen positive
* History of liver cirrhosis
* Persistently elevated liver transaminases, defined as ALT/AST at least 3 times the upper limit of normal for a minimum of 3 consecutive months
* Waitlisted for a multi-organ transplant
* Pregnant women
* Known allergy to sofosbuvir/velpatasvir
* Any condition, psychiatric or physical, that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study
* Ongoing therapy with amiodarone for atrial or ventricular arrhythmia Prescribed use of Amiodarone

Exclusion criteria (donors):

* Confirmed HIV positive (positive HIV-1 antibody, positive HIV-2 antibody, positive p24 antigen and/or positive HIV NAT)
* Confirmed HBV positive (positive hepatitis B surface antigen and/or HBV NAT) Known ongoing therapy for HCV

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 5 years
  Rate of adverse events due to sofosbuvir/velpatasvir (Epclusa) in patients in each experimental group
HCV free at 1 year | 1 year
  Proportion of participants in each experimental group who are free of HCV at 1 year following transplantation

SECONDARY OUTCOMES:
Transmission rate of HCV from HCVAb+/NAT- donors to HCVAb- recipients | 5 years
Incidence of allograft rejection | 5 years
Incidence of graft loss | 5 years
All-cause mortality | 5 years
Waitlist time after enrollment | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No